CLINICAL TRIAL: NCT00675623
Title: A Global Phase 3, Double-Blind, Placebo-Controlled Safety and Efficacy Study of Oral Dimebon in Patients With Mild-to-Moderate Alzheimer's Disease (CONNECTION)
Brief Title: A Safety and Efficacy Study of Oral Dimebon in Patients With Mild-To-Moderate Alzheimer's Disease
Acronym: CONNECTION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CONNECTION; DIM14
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease, clinical trial, memory loss, mitochondria,; investigational drug, neurodegenerative disease, dementia
MeSH Terms: conditions — Alzheimer Disease; Memory Disorders; Neurodegenerative Diseases; Dementia | interventions — latrepirdine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): Dimebon, 5 mg orally three times daily
  Interventions: Drug: Dimebon
- B (Experimental): Dimebon 20 mg orally three times daily
  Interventions: Drug: Dimebon
- C (Placebo Comparator): Placebo orally three times daily for six months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dimebon — Dimebon, 5 mg orally three times daily for six months
  Arms: A
Drug: Dimebon — Dimebon 20 mg orally three times daily for six months
  Arms: B
Drug: Placebo — Placebo three times daily for six months
  Arms: C

SUMMARY:
The Connection Study is a six-month confirmatory Phase 3 study to determine the safety and efficacy of Dimebon in the treatment of mild-to-moderate Alzheimer's disease (AD).

DETAILED DESCRIPTION:
This study is a randomized, placebo-controlled 6-month study designed as an adequate and well-controlled trial to demonstrate the safety and efficacy of Dimebon in the treatment of patients with mild-to-moderate AD. Dimebon is an investigational drug for Alzheimer's disease. The target of Dimebon's mechanism of action are the mitochondria (a cell's primary source of energy).The Connection Study is the second of two pivotal studies evaluating the effect of Dimebon. It is a 6-month study enrolling 525 patients in the United States, Europe, and South America. All patients completing the 6-month study will be eligible to receive Dimebon in an open-label extension trial.

The patient population will be carefully selected to ensure inclusion of patients with AD, rather than other types of dementia. Mild-to-moderate disease will be defined by the screening Mini-Mental State Examination (MMSE). Patients will attend study visits with caregivers who will provide information about the patient's condition.

ELIGIBILITY:
Inclusion Criteria:

* Mild-to-Moderate Alzheimer's disease
* Probable AD (National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) and Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV)
* MMSE score 10-24 inclusive
* Computerized tomography (CT) san or magnetic resonance imaging (MRI) consistent with AD
* Caregiver who cares for the patient at least 5 days per week

Exclusion Criteria:

* Anti-dementia drugs including cholinesterase-inhibitors or N-methyl-D-aspartate receptor (NMDA) receptor antagonists within 90 days
* Other causes of dementia
* Other primary psychiatric or neurological disorders
* Unstable medical illnesses or significant hepatic or renal disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To determine the effect of Dimebon as compared to placebo on the primary measure of cognition and memory, the Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog). | Week 26
To determine the effect of Dimebon as compared to placebo on the primary measure of global function, the Clinician's Interview-Based Impression of Change Plus Caregiver Input (CIBIC-plus). | Week 26

SECONDARY OUTCOMES:
To determine the effect of Dimebon as compared to placebo on a measure of self care and daily function, the Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL). | Week 26
To determine the effect of Dimebon as compared to placebo on a measure of behavior, the Neuropsychiatric Inventory (NPI). | Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Seely, MD, Study Director — Medivation, Inc.
Locations (28):
- United States (28):
  - Phoenix, Arizona
  - Costa Mesa, California
  - Fresno, California
  - Rancho Mirage, California
  - Hamden, Connecticut
  - New Haven, Connecticut
  - Norwalk, Connecticut
  - Hallandale, Florida
  - Hialeah, Florida
  - Miami, Florida
  - North Miami, Florida
  - Sunrise, Florida
  - West Palm Beach, Florida
  - Indianapolis, Indiana
  - Paducah, Kentucky
  - Newton, Massachusetts
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - Brooklyn, New York
  - Cedarhurst, New York
  - New York, New York
  - Rochester, New York
  - Staten Island, New York
  - Morganton, North Carolina
  - Centerville, Ohio
  - Norristown, Pennsylvania
  - Austin, Texas
  - Middleton, Wisconsin